CLINICAL TRIAL: NCT05672589
Title: To Compare Relaxed Rotational Thromboelastometry Cut-offs With Standard Cut-offs for Guiding Blood Product Use Before Invasive Procedures in Cirrhosis and Acute on Chronic Liver Failure Patients: A Randomized Controlled Trial
Brief Title: To Compare Relaxed Rotational Thromboelastometry Cut-offs With Standard Cut-offs for Guiding Blood Product Use Before Invasive Procedures in Cirrhosis and Acute on Chronic Liver Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-51
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-11

CONDITIONS: Liver Cirrhosis; Acute on Chronic Liver Failure
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxed rotational thromboelastometry (Experimental): Relaxed rotational thromboelastometry will be done 12 hr,24 hr,48 hr, 72 hr and if patients bleed.
  Interventions: Diagnostic Test: Relaxed Rotational Thromboelastometry
- Standard coagulation tests (Active Comparator): Standard coagulation tests will be done baseline,12 hr,24 hr,48 hr, 72 hr and if patients bleed
  Interventions: Diagnostic Test: Standard Coagulation Tests

INTERVENTIONS:
Diagnostic Test: Relaxed Rotational Thromboelastometry — Relaxed rotational thromboelastometry will be done 12 hr,24 hr,48 hr, 72 hr and if patients. bleed.
  Arms: Relaxed rotational thromboelastometry
Diagnostic Test: Standard Coagulation Tests — Standard coagulation tests will be done baseline,12 hr,24 hr,48 hr, 72 hr and if patients bleed.
  Arms: Standard coagulation tests

SUMMARY:
Hypothesis

Relaxed ROTEM cutoff guided blood product transfusion will result in less blood products use without increasing bleeding complications for invasive procedures in cirrhosis or acute on chronic liver failure (ACLF) patients

AIM:- To evaluate the efficacy and safety of Relaxed threshold (as compared to conventional thresholds) for blood product transfusion for invasive procedures in cirrhosis or acute on chronic liver failure (ACLF) patients

Objective -

Primary objective:

To compare the reduction in amount of total component transfused (ml/kg) in Relaxed Rotational Thromboelastometry based versus Conventional Rotational Thromboelastometry based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

Secondary objectives:

To compare the amount of FFP (ml/kg) transfused in Relaxed Rotational Thromboelastometry cut off based versus Standard Rotational Thromboelastometry cut off based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

To compare the amount of Platelet (ml/kg) transfused in Relaxed Rotational Thromboelastometry based versus Conventional Rotational Thromboelastometry based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

To compare the amount of cryoprecipitate (ml/kg) transfused in Relaxed Rotational Thromboelastometry based versus Conventional Rotational Thromboelastometry based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

To compare the bleeding rate in Relaxed Rotational Thromboelastometry cut off based versus Conventional Rotational Thromboelastometry cut off based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

To compare the rate of transfusion reactions in Relaxed Rotational Thromboelastometry based versus Conventional Rotational Thromboelastometry based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

To compare the cost incurred in Relaxed Rotational Thromboelastometry based versus Conventional Rotational Thromboelastometry based transfusion strategy in cirrhosis or acute on chronic liver failure (ACLF) patients.

DETAILED DESCRIPTION:
Methodology

Investigator will be following guidelines given by Society of Interventional Radiology for any intervention for coagulopathy correction.

Different procedures which are routinely carry out at our institute will be divided into high risk vs low risk as per Society of Interventional Radiology

Low risk: Peripherally inserted central catheter placement, Paracentesis, Thoracocentesis, Central venous cannulation, Lumbar puncture, Dialysis catheter placement

Low risk: Solid organ biopsies, Transjugular intrahepatic portosystemic shunts, Biliary interventions (cholecystostomy tube placement)

If the patient has evidence of ongoing sepsis (Positive blood culture, increased procalcitonin, shock, fever etc) or renal dysfunction, then he will be considered to be at high risk for the procedure.

After determining the risk category of the procedure, patients will decide to receive coagulopathy correction based on CCT (Society of Interventional Radiology). Those patients who do not require correction will be excluded.

For high risk procedures: PLT < 20, INR >2.5, Fibrinogen < 100 mg/dL

For low risk procedures: PLT < 30, INR > 2.0, Fibrinogen < 100 mg/dL

Those patients who will require coagulopathy correction will be randomized to receive correction based on standard ROTEM criteria versus Relaxed ROTEM criteria.

Standard ROTEM criteria:

CT EX >80 s �' FFP/PCC(if volume overload)

MCF EX <35 mm

MCF FIB <8 mm �' Cryoprecipitate transfusion

MCF FIB ≥8 mm �' Platelets transfusion

Relaxed ROTEM criteria:

CT EX >90 s �' FFP/PCC(if volume overload)

MCF EX <30 mm

MCF FIB <7 mm �' Cryoprecipitate transfusion

MCF FIB ≥7 mm �' Platelets transfusion

CCTs and/or ROTEM will be revised 12 hourly for 24 hours, then every 24 hours for next 48 hours; and if bleeding complications occur. However patients will undergo a procedure immediately after the coagulopathy correction based on baseline CCT and/or ROTEM. Patients will be followed up till day 28 post procedure for procedure related bleeding and non bleeding complications.

Acute kidney injury:

The Kidney Disease Improving Global Outcomes (KDIGO) guidelines define AKI as any of the following:

1. Increase in sCr by ≥0.3 mg/dl within 48 h or
2. Increase in sCr to ≥1.5x baseline, which is known or presumed to have occurred within the prior 7 days or
3. Urine volume <0.5 ml/kg/h for 6 h

Sepsis:

The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)

Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.

● Organ dysfunction can be identified as an acute change in total SOFA score ≥2 points consequent to the infection

Study population: All Cirrhosis and/or ACLF patients >18 yrs, scheduled to undergo an high risk invasive procedure with severe coagulopathy requiring correction as per risk category and degree of coagulopathy on conventional coagulation tests.

Study design: Randomized controlled trial

Study period: 1 years

Sample size: 1050

Assuming that the proportion of patients requiring any blood products transfusion (i.e either FFP/platelets/ cryoprecipitate), in standard criteria group: 20% [Ref:Pietri etal. HEPATOLOGY 2016;63:566-573] and Relaxed group criteria: 13% (1/3rd decrease).

Two-sided significance level(1-alpha): 95

Power(1-beta, % chance of detecting): 80

Ratio of sample size, Unexposed/Exposed: 1

Percent of Unexposed with Outcome: 20

Percent of Exposed with Outcome: 13

Investigator decided to enroll total 1050 patients considering 10% dropout rate, 525 subjects in each arm

Patients were randomized to either Relaxed ROTEM or conventional ROTEM transfusion groups in a 1:1 ratio by random computer generated sequence

Monitoring and assessment: All the parameters of the objective and also noted any adverse effects.

Stopping rule: If patient decided to withdraw from study

ELIGIBILITY:
Inclusion Criteria:

- All Cirrhosis and/or ACLF patients >18 yrs, scheduled to undergo an high risk invasive procedure with severe coagulopathy requiring correction as per risk category and degree of coagulopathy on conventional coagulation tests.

Exclusion Criteria:

1. Ongoing bleeding
2. Bleeding within last 3 days
3. ACLF patients going for LT may be added in exclusion criteria
4. Antiplatelet or anticoagulant therapy (discontinued <7 d before)
5. Hemodialysis in last 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the proportion of patients requiring any blood products transfusion (i.e FFP / platelets / cryoprecipitate) | 0 hours

SECONDARY OUTCOMES:
To compare the proportion of patients requiring FFP transfusion | 0 hours
To compare the proportion of patients requiring platelets transfusion | 0 hours
To compare the proportion of patients requiring cryoprecipitate transfusion | 0 hours
To compare the proportion of patients requiring tranexamic acid infusion | 0 hours
To compare the amount of FFP transfused (mL) in patients requiring FFP transfusion per patient | 0 hours
To compare the amount of platelets transfused (SDAP units) in patients requiring platelet transfusion per patient | 0 hours
To compare the amount of cryoprecipitate transfused (units) in patients requiring cryoprecipitate transfusion per patient | 0 hours
To compare the occurrence of bleeding, defined as overt bleeding or hemoglobin drop requiring transfusion with a target of 8 g/dL 28 days patient survival | 28 days
To compare the transfusion-related side effects, defined as any side effect occurring within 6 hours of blood products infusion; and Procedure-related complications other than bleeding | 6 hours
To compare the cost incurred | 0 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided